CLINICAL TRIAL: NCT01617252
Title: High Flow Nasal Oxygen Therapy for Hypoxemy After Cardiac Surgery
Acronym: Optiflow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BRD/10/09-H
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Hypoxemic Acute Respiratory Failure
Keywords: Cardiac surgery; Acute respiratory failure; High flow oxygen therapy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optiflow (Experimental)
  Interventions: Device: Optiflow / Facial mask
- Facial mask (Experimental)
  Interventions: Device: Optiflow / Facial mask

INTERVENTIONS:
Device: Optiflow / Facial mask — J0: randomization (Optiflow® or facial mask), lung X-ray, kinesiotherapy H0 : clinical examination, blood gas, respiratory frequency H1 : clinical examination, blood gas, respiratory frequency H6 : clinical examination, blood gas J1: clinical examination, blood gas, respiratory frequency, lung X-ray, diaphragmatic echography, kinesiotherapy J2: clinical examination, blood gas, lung X-ray, kinesiotherapy Follow-up (until withdrawal of Optiflow or facial mask): clinical examination, blood gas, lung X-ray, kinesiotherapy

SUMMARY:
The main objective of this study is to evaluate the gas exchange (ventilation-perfusion ratio) with the system Optiflow® compared to facial mask among patients having an acute respiratory failure after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication of coronary artery bypass
* Absence of preoperative respiratory failure
* Hypoxia after extubation defined as SpO2 < 96% with Venturi mask 50% 8L/min
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Patients requiring an imminent intubation, in coma or respiratory exhaustion, in a state of shock or severe rhythm disorders
* Hemodynamic instability, low flow rate
* Pneumothorax or hemothorax
* Bleeding major, ischemic signs
* Ventricular arrhythmia
* Respiratory failure
* Non controlled hyperalgia
* Alteration of mental status
* Cardiac surgery patients in post-operative valve surgery associated with coronary artery bypass surgery or isolated valve surgery
* Pregnancy
* Major under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Measure of PaO2/FiO2 ratio | One hour and 24 hours
  The main objective of this study is to evaluate the gas exchange (ventilation-perfusion ratio) with the system Optiflow® compared to facial mask among patients having an acute respiratory failure after cardiac surgery.

SECONDARY OUTCOMES:
Scale of satisfaction completed by the patient | at withdrawal of oxygen system
  To evaluate the tolerance of high flow oxygen therapy: satisfaction scale
Measure of pH, SatO2, PaO2, FiO2 | 2 days
  To evaluate hypoxia duration
Number of days of hospitalization | at day 28
  To evaluate the duration of hospitalization with the medical device
Measure of PCO2 and respiratory frequency | One day
  To evaluate PCO2 and respiratory frequency at H+1 and J1
Possibility of patient transfer in conventional service | at day 5
  To evaluate the reception in post reanimation if transfer under oxygen therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France